CLINICAL TRIAL: NCT05638620
Title: Evaluating the Effectiveness of Dual Sympathetic Blocks for Patients Experiencing Sympathetically-Mediated Symptoms From Post-Acute Sequelae of SARS-CoV-2 (PASC)
Brief Title: Dual Sympathetic Blocks for Patients Experiencing Sympathetically-Mediated Symptoms From Long COVID
Acronym: DSBLongCOVID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonathann Kuo, MD (Other)
Responsible Party: Sponsor-Investigator, Jonathann Kuo, MD, Medical Director, Hudson Medical
Organization: Hudson Medical (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRANY # 22-02-733-993
Record Dates: First submitted 2022-11-22; First posted 2022-12-06 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Post Acute COVID-19 Syndrome; Long COVID; Long Covid19; COVID-19 Recurrent; Post-Acute COVID-19; Post-Acute COVID-19 Infection; SARS-CoV2 Infection; Post Acute Sequelae of COVID-19; Dysautonomia; Dysautonomia Like Disorder; Dysautonomia Orthostatic Hypotension Syndrome; Post COVID-19 Condition; Post-COVID Syndrome; Post COVID-19 Condition, Unspecified; Post-COVID-19 Syndrome
Keywords: COVID; long covid; SARS-COV2; COVID-19; long COVID-19; post covid; dysautonomia; stellate ganglion block; dual sympathetic block; SGB; DSB
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Autonomic Nervous System Diseases; Dysautonomia like disorder; Shy-Drager Syndrome | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This will be a single-site, non-randomized, open-label, prospective study to evaluate the effects of bilateral Dual Sympathetic Blocks (DSB) on the dysautonomic symptomatology of Post-Acute Sequelae of SARS-CoV-2 (PASC). Patients will be evaluated for pain interference and dysautonomic symptomatology by the PROMIS-29 and COMPASS-31 scores at 0,1, and 4 weeks.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Active (Experimental): This is a non-randomized, non-blinded study. Participants eligible for this study will receive active treatment. Dual Sympathetic Blocks of the stellate ganglion are minimally- invasive outpatient procedures performed under monitored care anesthesia (light sedation). Under ultrasound visualization, a small needle is guided into the neck region that contains the stellate ganglion nerve cluster at C6-C7. Once the needle position is confirmed, a local anesthetic (7 cc of 0.5% bupivacaine/Marcaine) is injected around the stellate ganglion by the Principal Investigator. This procedure is repeated at the C3-C4 level to block the superior cervical ganglion nerve cluster (3 cc of 0.5% bupivacaine/Marcaine).
  Interventions: Drug: stellate ganglion block with 0.5% bupivacaine

INTERVENTIONS:
Drug: stellate ganglion block with 0.5% bupivacaine — The stellate ganglion block is being done on both sides of the neck. The stellate ganglion block will be performed on the right side at the first visit. The procedure will be repeated on the left side one week after the first injection.
  This study is not intended to be reported to FDA as a well-controlled study in support of a new indication for use nor intended to be used to support any other significant change in the labeling for the drug. Similar to a phase 1 clinical trial, the main purpose of this study is to gather data and assess changes in patient-reported outcomes with the stellate ganglion blocks as treatment for their sympathetically-mediated long COVID symptoms. As a general rule, phase 1 studies require a low number of patients, typically 12-20 subjects. There is considerable uncertainty regarding long COVID as a disease state, so data from even small numbers of patients in a well-designed clinical trial will make steps towards reducing that uncertainty.
  Other Names: Dual Sympathetic Block; Stellate ganglion nerve block

SUMMARY:
The main purpose of this study is to gather data and assess changes in patient-reported outcomes with the stellate ganglion blocks as treatment for their sympathetically-mediated long COVID symptoms.

DETAILED DESCRIPTION:
1.1 Background 1.1.1.Post-Acute Sequelae of SARS-CoV-2 (PASC) Since the onset of the COVID-19 pandemic, demands for rapid mobilization of research initiatives and treatment protocols continue to grow. While some people recover quickly from COVID-19, an increasing number of individuals previously infected with the SARS-CoV-2 virus report experiencing new, returning, or ongoing health problems long after recovery from the acute disease.The CDC and NIH define these long-term effects of COVID-19 by the broad research term Post-Acute Sequelae of SARS-CoV-2 infection (PASC), which is characterized by the presence of persistent or recurrent symptoms in patients who have recovered from an acute SARS-CoV-2 infection. PASC, also known as post-COVID conditions (PCC) or long COVID, presents in different ways and can affect the function of many different organs and systems including respiratory, neurological, and digestive systems. Most commonly, PASC symptoms include fatigue, post-exertional malaise, shortness of breath, "brain fog," sleep problems, fever, anxiety, and depression. Other symptoms include persistent cough, chest pain or chest discomfort, headache, heart palpitations, joint or muscle pain, diarrhea, nausea, abdominal pain, fever, dizziness, anosmia, or ageusia. Symptoms can vary between patients as some will experience only one of these symptoms while others may have two or more. The severity of symptoms range from mild to severe and can be debilitating. There is no test to diagnose post-COVID conditions. The symptoms of PASC can be difficult to explain and clinical evaluations or testing from routine blood tests, chest x- rays, and electrocardiograms may be normal, making it difficult for healthcare providers to recognize. Though more prevalent in people who had severe COVID-19 illness, anyone who has been infected with the virus that causes COVID-19 can experience post-COVID conditions, even people who had mild illness or no symptoms from a SARS- CoV-2 infection. Healthcare providers consider a diagnosis of post-COVID conditions based on a patient's health history, including if they had a diagnosis of COVID-19 either by a positive test or by symptoms or exposure. PASC can have significant effects beyond managing the physical symptoms. Many people report that long COVID symptoms prevent them from returning to work or school or cause them difficulties in performing everyday tasks or even walking short distances. Pain centers seeing patients with PASC report most patients would meet the definition of chronic primary pain with major distress based on the ICD-11 chapter for chronic pain (Wadehra). Furthermore, recent guidance states PASC, or Long COVID, can qualify as a disability under the American Disability Act if it limits at least one major life activity. The current research and understanding of PASC indicates it acts similarly to syndromes of chronic pain and sympathetic nervous system dysfunction that may be targeted by existing interventions. The symptoms can be functionally debilitating and can severely diminish quality of life, so identifying effective treatments and management strategies that address this disease may prove to have significant implications in the wake of the COVID-19 Pandemic.

1.1.2. Treatment for Post-Acute Sequelae of SARS-CoV-2 (PASC) As PASC has only recently been defined as a distinct disease state, it is not well understood yet and targeted and effective treatment options are extremely limited. PASC can affect many different organ systems, so current treatments are often multi- disciplinary, focusing on symptomatic management and treatment of underlying health problems. Clinicians have suggested that effective treatment should manage related pain and dysfunction. Many PASC symptoms that fail to respond to traditional treatment protocols are associated with dysautonomia. Dysautonomia is abnormal activity of involuntary body functions that are regulated by the sympathetic nervous system, such as heart rate, breathing and digestion. Sympathetic innervation plays a vital role in the communication between the immune system and the nervous system, but pathologies, such as elevated cytokine levels, can disrupt this relationship and promote sympathetic responses and subsequent inflammatory problems. In this way, the well-documented cytokine storm response to a SARS-CoV-2 infection results from sympathetic activation as the autonomic nervous system responds to pro-inflammatory cytokines. During elevated sympathetic signaling, the brainstem responds by integrating this information into "sickness behaviors," a set of behavioral responses which closely resembles PASC symptoms. As PASC may persist over weeks or months, persistent dysfunctional or inappropriate sympathetic signaling may potentially contribute to or exacerbate symptoms. Furthermore, prolonged dysautonomia is associated with impaired cerebral blood flow (CBF) in conditions such as myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS), postural orthostatic tachycardia syndrome (POTS), and other poorly understood sympathetically-mediated chronic illnesses like complex regional pain syndrome (CRPS). In general, impaired CBF causes a range of clinical symptoms such as cognitive dysfunction, impaired memory and attention, and reduced visual, gustatory or olfactory function. The clinical presentations in these conditions parallel many common symptoms of PASC. Ongoing research and case studies are working to better understand the pathophysiology and effective treatments for PASC. The purpose of this study is to identify patients with continued hyperactivation of the sympathetic nervous system that can be targeted with existing treatments. A cases series conducted in 2021 showed promising results supporting Stellate ganglion blocks to reduce symptoms of Long COVID, or PASC. The case series reported sustained positive clinical outcomes for two Long COVID patients after treatment with SGB, identifying the pathophysiology for their symptoms as a regional sympathetically mediated dysautonomia. The results suggest SGB could be an effective intervention for at least a subset of Long COVID patients. Researchers conclude that although the application of SGB in PASC is novel, it is a promising and attractive therapeutic for a condition that currently lacks effective treatment options.

1.1.3. Dual Sympathetic Blocks (Stellate Ganglion Blocks) Sympathetic nerve blocks are established procedures used by many pain management providers as an effective method to diagnose or treat pain involving the nerves of the sympathetic nervous system. A block of the sympathetic nerves at the Stellate Ganglion in the upper neck has been used for decades to treat complex, sympathetically-mediated pain syndromes affecting the head, face, neck and arms. The stellate ganglion nerve bundle carries sympathetic signaling to many body regions and organs, including the head, neck, upper limbs, thymus, heart, lungs, lacrimal gland, salivary gland, thyroid gland and pineal gland. Injection of local anesthetic near the stellate ganglion can block activity of the entire cervical sympathetic chain, as evidenced by the physiological signs of a successful stellate ganglion block (SGB) collectively known as "Horner's Syndrome" which includes ipsilateral ptosis, meiosis, anhidrosis, and facial flushing. Researchers suggest the SGB can alleviate symptoms of dysautonomia by providing local recalibration of regional sympathetic influence, central integration of the effects of increased CBF, or rebalancing of the interaction between the nervous and immune systems. During the procedure, a physician uses x-ray or ultrasound imaging to guide a needle into a bundle of nerves located near the base of the neck. The physician then injects a local anesthetic into the nerve tissue like a dentist delivers numbing medicine before a dental procedure. The anesthetic lasts only a few hours, but the effects of the procedure can last for several weeks or longer in some cases. The use of Marcaine (bupivacaine) is indicated for local or regional anesthesia or analgesia for surgery, dental and oral surgery procedures, diagnostic and therapeutic procedures (including sympathetic nerve blocks), and for obstetrical procedures. The drug is lawfully marketed as a prescription drug product, and this investigation is not intended to support a significant change in the advertising for the product. There is increasing evidence that PASC has a similar profile to many pain syndromes, and dysautonomia appears to play an important role among the clinical manifestations in both the acute and chronic phase of SARS-CoV-2 infection. Thus, the use of sympathetic blocks in this study is meant to be included under the current indications for the treatment: an effective method to diagnose or treat pain involving the nerves of the sympathetic nervous system.

1.1.4. Theoretical Models There are a few published case series that seek to make further connections between PASC symptoms and autonomic dysfunction. Researchers express that the safety profile for Dual Sympathetic Blocks (Stellate ganglion blocks) is well established and has been used for nearly a century to treat a variety of sympathetically-mediated medical conditions. The lack of effective treatments for Long COVID/PASC makes the DSB an attractive therapeutic modality that deserves further investigation.

1.2 Rationale for Current Study This investigation is not intended to be reported to FDA as a well-controlled study in support of a new indication for use nor intended to be used to support any other significant change in the labeling for the drug. Clinicians have suggested that effective treatment for PASC should manage related pain and dysfunction. A sympathetic nerve block is used to both diagnose dysfunction and treat pain caused by the sympathetic nervous system. Sympathetic nerve blocks including the stellate ganglion blocks have been widely used by pain management physicians and their safety is well proven for the treatment of sympathetically-mediated pain syndromes.

Though PASC has only recently been defined, emerging and continued research supports the understanding that the SARS-CoV-2 infection affects the autonomic nervous system. Therefore, this study hopes to analyze the effectiveness of sympathetic nerve blocks to identify and treat symptoms of sympathetically-mediated pain or dysfunction in patients with PASC. The propensity of the PASC to lead to long-term illness and impairments calls for clinical trials aimed at prevention and treatment. The PROMIS-29 and COMPASS-31 surveys will be administered as part of the screening process to identify autonomic dysfunction. Patients who report symptoms of pain that interferes with daily function and at least one autonomic symptom that recurs or persists for 4 weeks or more after a SARS-CoV-2 infection meet the current criteria for PASC and may be eligible to participate. Findings from the current study may provide much needed insight into the state of the PASC disease and guidance for future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Prior confirmed COVID-19 diagnosis by standard RT-PCR assay or equivalent testing
* Persistent symptoms that continue four or more weeks after the start of a COVID-19 infection
* Quantified autonomic symptoms from at least one domain as reported by the patient on the screener Composite Autonomic Symptom Score (COMPASS-31). The COMPASS-31 assesses 6 domains of autonomic symptoms: Orthostatic Intolerance, Vasomotor, Secretomotor, Gastrointestinal, Bladder, and Pupillomotor.
* Quantified pain symptoms of pain interference or pain intensity as reported by the patient on the screener Patient-Reported Outcomes Measurement Information System (PROMIS-29)

Exclusion Criteria:

* Under age 18
* Prior SGB
* Allergy to amide local anesthetics (e.g., ropivacaine, bupivacaine/Marcaine)
* Pregnancy
* Current anticoagulant use
* History of a bleeding disorder
* History of glaucoma
* Infection or mass at injection site
* For the consistency of this study, patients who deny all autonomic symptoms on the COMPASS-31 or pain symptoms on the PROMIS-29 will also be excluded

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes: PROMIS-29 Score | 1 month
  The primary objective of the clinical effectiveness trial is to evaluate whether Dual Sympathetic Blocks performed at 0 and 1 weeks will improve patient-reported outcomes of depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities status. These domains are measured as reflected by Patient-Reported Outcomes Measurement Information System (PROMIS-29) total scores between baseline and 4 weeks
Depression | 1 month
  PROMIS-29 survey will measure changes in each domain scores between baseline and 4 weeks.
Anxiety | 1 month
  PROMIS-29 survey will measure changes in each domain scores between baseline and 4 weeks.
Physical function | 1 month
  PROMIS-29 survey will measure changes in each domain scores between baseline and 4 weeks.
Pain interference | 1 month
  PROMIS-29 survey will measure changes in each domain scores between baseline and 4 weeks.
Fatigue | 1 month
  PROMIS-29 survey will measure changes in each domain scores between baseline and 4 weeks.
Sleep disturbance | 1 month
  PROMIS-29 survey will measure changes in each domain scores between baseline and 4 weeks.
Ability to participate in social roles and activities status | 1 month
  PROMIS-29 survey will measure changes in each domain scores between baseline and 4 weeks.

SECONDARY OUTCOMES:
Autonomic Symptoms: COMPASS-31 Score | 1 month
  The secondary objective of the clinical effectiveness trial is to evaluate whether Dual Sympathetic Blocks performed at 0 and 1 weeks will improve Dysautonomia symptoms as reflected by corresponding Composite Autonomic Symptom Scale 31 (COMPASS-31) scores between baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathann Kuo, MD, Principal Investigator — Medical Director
Locations (1):
- Hudson Medical, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
All information will be kept confidential. Study-related information will be stored securely at the study site. All participant information will be stored with limited access. All reports, data collection, and administrative forms will be identified by a coded ID [identification] number only to maintain participant confidentiality. Records that contain names or other personal identifiers, such as locator forms and informed consent forms, will be stored separately from study records identified by code number. All local databases will be secured with password-protected access systems. Forms, lists, logbooks, appointment books, and any other listings that link participant ID numbers to other identifying information will be stored in a separate, locked file with limited access.

REFERENCES:
- [Background] Attal N, Martinez V, Bouhassira D. Potential for increased prevalence of neuropathic pain after the COVID-19 pandemic. Pain Rep. 2021 Jan 27;6(1):e884. doi: 10.1097/PR9.0000000000000884. eCollection 2021 Jan-Feb. PMID 33537521
- [Background] Bucsek MJ, Giridharan T, MacDonald CR, Hylander BL, Repasky EA. An overview of the role of sympathetic regulation of immune responses in infectious disease and autoimmunity. Int J Hyperthermia. 2018 Mar;34(2):135-143. doi: 10.1080/02656736.2017.1411621. PMID 29498310
- [Background] Carmona-Torre F, Minguez-Olaondo A, Lopez-Bravo A, Tijero B, Grozeva V, Walcker M, Azkune-Galparsoro H, Lopez de Munain A, Alcaide AB, Quiroga J, Del Pozo JL, Gomez-Esteban JC. Dysautonomia in COVID-19 Patients: A Narrative Review on Clinical Course, Diagnostic and Therapeutic Strategies. Front Neurol. 2022 May 27;13:886609. doi: 10.3389/fneur.2022.886609. eCollection 2022. PMID 35720084
- [Background] Carod-Artal FJ. Infectious diseases causing autonomic dysfunction. Clin Auton Res. 2018 Feb;28(1):67-81. doi: 10.1007/s10286-017-0452-4. Epub 2017 Jul 20. PMID 28730326
- [Background] Dani M, Dirksen A, Taraborrelli P, Torocastro M, Panagopoulos D, Sutton R, Lim PB. Autonomic dysfunction in 'long COVID': rationale, physiology and management strategies. Clin Med (Lond). 2021 Jan;21(1):e63-e67. doi: 10.7861/clinmed.2020-0896. Epub 2020 Nov 26. PMID 33243837
- [Background] Datta R, Agrawal J, Sharma A, Rathore VS, Datta S. A study of the efficacy of stellate ganglion blocks in complex regional pain syndromes of the upper body. J Anaesthesiol Clin Pharmacol. 2017 Oct-Dec;33(4):534-540. doi: 10.4103/joacp.JOACP_326_16. PMID 29416250
- [Background] Ganesh R, Ghosh AK, Nyman MA, Croghan IT, Grach SL, Anstine CV, Salonen BR, Hurt RT. PROMIS Scales for Assessment of Persistent Post-COVID Symptoms: A Cross Sectional Study. J Prim Care Community Health. 2021 Jan-Dec;12:21501327211030413. doi: 10.1177/21501327211030413. PMID 34231395
- [Background] Goodman BP, Khoury JA, Blair JE, Grill MF. COVID-19 Dysautonomia. Front Neurol. 2021 Apr 13;12:624968. doi: 10.3389/fneur.2021.624968. eCollection 2021. PMID 33927679
- [Background] Grebe KM, Takeda K, Hickman HD, Bailey AL, Embry AC, Bennink JR, Yewdell JW. Cutting edge: Sympathetic nervous system increases proinflammatory cytokines and exacerbates influenza A virus pathogenesis. J Immunol. 2010 Jan 15;184(2):540-4. doi: 10.4049/jimmunol.0903395. Epub 2009 Dec 16. PMID 20018617
- [Background] Kang CK, Oh ST, Chung RK, Lee H, Park CA, Kim YB, Yoo JH, Kim DY, Cho ZH. Effect of stellate ganglion block on the cerebrovascular system: magnetic resonance angiography study. Anesthesiology. 2010 Oct;113(4):936-44. doi: 10.1097/ALN.0b013e3181ec63f5. PMID 20823762
- [Background] Kenney MJ, Ganta CK. Autonomic nervous system and immune system interactions. Compr Physiol. 2014 Jul;4(3):1177-200. doi: 10.1002/cphy.c130051. PMID 24944034
- [Background] Liu LD, Duricka DL. Stellate ganglion block reduces symptoms of Long COVID: A case series. J Neuroimmunol. 2022 Jan 15;362:577784. doi: 10.1016/j.jneuroim.2021.577784. Epub 2021 Dec 8. PMID 34922127
- [Background] Lipov EG, Navaie M, Brown PR, Hickey AH, Stedje-Larsen ET, McLay RN. Stellate ganglion block improves refractory post-traumatic stress disorder and associated memory dysfunction: a case report and systematic literature review. Mil Med. 2013 Feb;178(2):e260-4. doi: 10.7205/MILMED-D-12-00290. PMID 23764335
- [Background] Moon HS, Chon JY, Lee SH, Ju YM, Sung CH. Long-term Results of Stellate Ganglion Block in Patients with Olfactory Dysfunction. Korean J Pain. 2013 Jan;26(1):57-61. doi: 10.3344/kjp.2013.26.1.57. Epub 2013 Jan 4. PMID 23342209
- [Background] Park HM, Kim TW, Choi HG, Yoon KB, Yoon DM. The change in regional cerebral oxygen saturation after stellate ganglion block. Korean J Pain. 2010 Jun;23(2):142-6. doi: 10.3344/kjp.2010.23.2.142. Epub 2010 May 31. PMID 20556217
- [Background] Pongratz G, Straub RH. The sympathetic nervous response in inflammation. Arthritis Res Ther. 2014;16(6):504. doi: 10.1186/s13075-014-0504-2. PMID 25789375
- [Background] Qin Y, Wu J, Chen T, Li J, Zhang G, Wu D, Zhou Y, Zheng N, Cai A, Ning Q, Manyande A, Xu F, Wang J, Zhu W. Long-term microstructure and cerebral blood flow changes in patients recovered from COVID-19 without neurological manifestations. J Clin Invest. 2021 Apr 15;131(8):e147329. doi: 10.1172/JCI147329. PMID 33630760
- [Background] Raveendran AV, Jayadevan R, Sashidharan S. Long COVID: An overview. Diabetes Metab Syndr. 2021 May-Jun;15(3):869-875. doi: 10.1016/j.dsx.2021.04.007. Epub 2021 Apr 20. PMID 33892403
- [Background] Rae Olmsted KL, Bartoszek M, Mulvaney S, McLean B, Turabi A, Young R, Kim E, Vandermaas-Peeler R, Morgan JK, Constantinescu O, Kane S, Nguyen C, Hirsch S, Munoz B, Wallace D, Croxford J, Lynch JH, White R, Walters BB. Effect of Stellate Ganglion Block Treatment on Posttraumatic Stress Disorder Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):130-138. doi: 10.1001/jamapsychiatry.2019.3474. PMID 31693083
- [Background] Scala I, Bellavia S, Luigetti M, Brunetti V, Broccolini A, Gabrielli M, Zileri Dal Verme L, Calabresi P, Della Marca G, Frisullo G. Autonomic dysfunction in non-critically ill COVID-19 patients during the acute phase of disease: an observational, cross-sectional study. Neurol Sci. 2022 Aug;43(8):4635-4643. doi: 10.1007/s10072-022-06136-2. Epub 2022 May 24. PMID 35608736
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] Tian T, Wu J, Chen T, Li J, Yan S, Zhou Y, Peng X, Li Y, Zheng N, Cai A, Ning Q, Xiang H, Xu F, Qin Y, Zhu W, Wang J. Long-term follow-up of dynamic brain changes in patients recovered from COVID-19 without neurological manifestations. JCI Insight. 2022 Feb 22;7(4):e155827. doi: 10.1172/jci.insight.155827. PMID 35191397
- [Background] Tian Y, Wittwer ED, Kapa S, McLeod CJ, Xiao P, Noseworthy PA, Mulpuru SK, Deshmukh AJ, Lee HC, Ackerman MJ, Asirvatham SJ, Munger TM, Liu XP, Friedman PA, Cha YM. Effective Use of Percutaneous Stellate Ganglion Blockade in Patients With Electrical Storm. Circ Arrhythm Electrophysiol. 2019 Sep;12(9):e007118. doi: 10.1161/CIRCEP.118.007118. Epub 2019 Sep 13. PMID 31514529
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Umeyama T, Kugimiya T, Ogawa T, Kandori Y, Ishizuka A, Hanaoka K. Changes in cerebral blood flow estimated after stellate ganglion block by single photon emission computed tomography. J Auton Nerv Syst. 1995 Jan 3;50(3):339-46. doi: 10.1016/0165-1838(94)00105-s. PMID 7714328
- [Background] Vallee A. Dysautonomia and Implications for Anosmia in Long COVID-19 Disease. J Clin Med. 2021 Nov 25;10(23):5514. doi: 10.3390/jcm10235514. PMID 34884216
- [Background] Wadehra S. COVID Long Haulers and the New Chronic Pain Profile . Pract Pain Manag. 2022;22(1).
- [Background] Wulf H, Maier C. [Complications and side effects of stellate ganglion blockade. Results of a questionnaire survey]. Anaesthesist. 1992 Mar;41(3):146-51. German. PMID 1570888
- See also: Stellate Ganglion Block (SGB) for COVID-19 Acute Respiratory Distress Syndrome (ARDS). ClinicaTrials.gov identifier NCT04402840. Updated November 3, 2020. Accessed October 11, 2022. — https://clinicaltrials.gov/ct2/show/NCT04402840